CLINICAL TRIAL: NCT06195111
Title: A Real-world Study of Trifluridine/Tipiracil Containing Regimen for the Treatment of Patients With Metastatic Colorectal Cancer (REFLECT Study)
Brief Title: A Real-world Study of Trifluridine/Tipiracil Containing Regimen for the Treatment of Patients With mCRC (REFLECT Study)
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0994
Record Dates: First submitted 2023-12-24; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trifluridine/Tipiracil: Patients with metastatic colorectal cancer plan to recieve Trifluridine/Tipiracil-containing treatment will be enrolled in this study. The prescription all determined by doctor based on patient's situation.
  Interventions: Drug: Trifluridine/Tipiracil

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — This a rospective observational study. There is no treatment allocation. Patients administered Trifluridine/Tipiracil by prescription
  Other Names: TAS-102; FTD/TPI; Lonsurf

SUMMARY:
A real-world study of trifluridine/tipiracil containing regimen for the treatment of patients with metastatic colorectal cancer. A total of 200 patients planned to be enrolled.

DETAILED DESCRIPTION:
This is a non-randomized, uncontrolled, multicenter real-world study. The total number of subjects is 200. The objective is to observe and evaluate the efficacy and safety of Trifluridine/Tipiracil alone or in combination with other therapies in the treatment of metastatic colorectal cancer in real-world environment. The primary endpoints is Progression-free survival (PFS). Secondary endpoints are overall survival (OS), Objective response rate(ORR), Disease control rate(DCR), progression-free survival (PFS), and Quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to fulfill all of the following criteria at enrollment:

* Male and female patients with ≥18 years of age;
* Patients with metastatic colorectal cancer confirmed by histopathology;
* Be willing to use reliable contraceptive methods and refrain from sperm donation throughout the study period and within 3 months after the last dose;
* Voluntarily join the study and provide written informed consent to participate in the study;
* Have traceable medical history during the treatment;
* Doctor believe the patients can benefit from the study.

Exclusion Criteria:

Patients fulfilling any of the following criteria at enrollment are not eligible for inclusion in this study:

* Failure to sign informed consent;
* Patients with contraindications to Trifluridine/Tipiracil;
* Female subjects who have a positive pregnancy test or are breastfeeding;
* Any medical or psychological condition in the treating physician's opinion which may prevent the patient from the study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, being treated for mCRC with Trifluridine/Tipiracil-containing regimen.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-free survival) | Approximately 12 months
  Progression-free survival defined as the time elapsed between the randomization and the date of radiologic tumour progression according to RECIST version 1.1 by investigator's judgement or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
OS (Overall Survival) | Approximately 12 months
  Overall survival defined as the observed time elapsed between the date of first treatment and the date of death due to any cause.
ORR（Objective response rate） | Approximately 12 months
  Objective Response Rate defined as the proportion of patients with objective evidence of complete response (CR) or partial response (PR) according to RECIST version 1.1 criteria and using investigator's tumor assessment.
DCR (Disease control rate) | Approximately 12 months
  Disease control rate defined as the proportion of patients with objective evidence of CR or PR or stable disease (SD) according to RECIST version 1.1 criteria and using investigator's tumor assessment.
Quality of life: EORTC QLQ-C30 | Approximately 12 months
  Assess patients health and activities using the European Organization for Research and Treatment of Cancer Core Quality of Life (EORTC QLQ-C30) module.

IPD SHARING:
Plan to Share IPD: No